CLINICAL TRIAL: NCT00755521
Title: Study Proposal - A Randomized Double-blinded Study Comparing Adding Etoricoxib Versus Placebo to Female Patients With Fibromyalgia-analysis of Organic and Psychiatric Measures
Brief Title: Study Assessing the Efficacy of Etoricoxib in Female Patients With Fibromyalgia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0134-08-MMC
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; tenderness; widespread pain; comrbidity
MeSH Terms: conditions — Fibromyalgia | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (No Intervention)
- A (Experimental): adding Etoricoxib to the basic therapeutic regimen
  Interventions: Drug: etoricoxib

INTERVENTIONS:
Drug: etoricoxib — Treating Fibromyalgia with etoricoxib
  etoricoxib - 90mg
  Other Names: Arcoxia
  Arms: A

SUMMARY:
The main of the proposed study is to assess whether the use of the Cox-2 inhibitor Etoricoxib is beneficial for the use in fibromyalgia. We intend to seek whether this medication may improve psychiatric and rheumatologic parameters of the disease.

DETAILED DESCRIPTION:
The fibromyalgia syndrome (FMS) is an ill-defined clinical disorder characterized by widespread pain and diffuse tenderness which is assessed at specified anatomical locations. The FMS is 10 times more common in females, and its prevalence in the community increases from two percent at age 20 to eight percent at age 70. Although the American College of Rheumatology (ACR) has defined classification criteria for the diagnosis of the FMS its' pathogenesis remains vague. Diffuse and persistent musculoskeletal pain, consistent with the mentioned ACR criteria have also been reported among patients with other ill defined medical conditions such as migraines, chronic fatigue pain, myofascial pain, irritable bowel syndrome which presentation often overlaps with the FMS.

There are mounting data supporting an overlap between the FMS and psychiatric conditions including depression, panic disorders and anxiety. For example, a lifetime history of major depression has been reported in 50% to 70% of patients with FMS and current depression was detected in 18% to 36% of patients with the FMS. This association has been questioned raising the possibility that this high prevalence reflects the long term outcome of coping with chronic disabling pain and disability.

Anti-depressants are the corner stone of therapy in FMS. Benzodiazepines and recent experience with melatonin has been implicated in order to alleviate sleep disturbances that are so often encountered among patients with this disorder. Nevertheless, patients with the FMS often need therapeutical medications in order to ease acute exacerbations of diffuse pain which are often provoked by mental or physical stressors.

Non-steroidal anti-inflammatory drugs (NSAIDs), COX-2-selective agents and acetaminophen are often used by a large number of FMS patients seeking a relief of acute pain. However, numerous studies have failed to confirm their effectiveness as analgesics in FMS, although there is limited evidence that patients may experience enhanced analgesia when treated with combinations of NSAIDs and other agents.

We believe that successful relief of diffuse pain may sever the bond tying pain and increased anxiety which is so characteristic in these patients. Furthermore, a clinical path that underlines the importance of pain relief may ensure the adherence and compliance that are needed to other elements of the therapeutical multidimensional approach in FMS and may be even improve psychiatric comorbidity that stem from the chronic non relenting pain.

A major factor limiting use of NSAIDs is concern for the development of gastrointestinal complications such as bleeding. COX-2 selective inhibitors were developed to decrease the risk of gastrointestinal tract injury and to avoid the anti-platelet effect of traditional NSAIDs. The recent MEDAL study has confirmed this finding by randomizing more than 30,000 patients to either etoricoxib or to the traditional NSAID diclofenate. Furthermore, the MEDAL investigators demonstrated similar cardiovascular outcome measures in both patient groups showing that the use of this has a similar cardiovascular safety profile as the traditional used NSAIDS. Using a safe analgesic with a low rate of adverse events in FMS patients, a population with enhanced somatoform ideation, is of great importance and may also insure the adherence to the other components of therapy.

Hypothesis - Adding etoricoxib, a COX-2 selective inhibitor, to the therapeutic regimens of patients with the FMS may ease their degree of pain; improve measures of over all quality of life, disability, sleep, anxiety and depression.

Objectives - Organic, mental and functional aspects of the FMS will be assessed in patients treated with etoricoxib (as an "add on") compared to placebo. The protocol-defined primary outcome measure will be pain severity as measured by the self-reported BPI (short form) average pain severity score (15).

Secondary endpoints will include tender point count, validated parameters that measure quality of life, quality of sleep, disability, pain, depression and anxiety and the fibromyalgia impact questionnaire (which measures physical function, pain assessment, fatigue and distress). The study will include eighty patients.

ELIGIBILITY:
Inclusion Criteria:

* • Women with established primary FMS who signed an informed consent form

  * Women 18-75 years old.
  * The score on the average pain severity item of the BPI is > 5 at randomization.
  * Patients on stable physical therapy or anelgestic pain treatment throughout the duration of the study.

Exclusion Criteria:

* • Confirmed pregnancy

  * Breast feeding patients
  * Patients with active coronary artery disease with documented myocardial ischemia proven by coronary angiography, thallium scan or exercise stress test.
  * Patients with congestive heart failure
  * Patients with coexistent neoplastic conditions (not including basal cell carcinoma)
  * Patients with coexistent t rheumatic/inflammatory conditions
  * Patients with active gastrointestinal bleeding
  * Patients with renal failure
  * Patients with comorbid conditions causing significant disability
  * Patients with uncontrolled hypertension.
  * Patient with contraindications for the trial drug based on the drug's physician leaflet.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-10 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Brief pain inventory | 6 weeks

SECONDARY OUTCOMES:
Tender point count, SF-36, Mini International Neuropsychiatric Interview | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Howard Amital, MD MHA, Principal Investigator — Meir Medical Center
Locations (1):
- Department of Medicine 'D', Meir Medical Center, Kfar Saba, Israel